CLINICAL TRIAL: NCT01545479
Title: Renal Oxygen Content is Increased in Healthy Subjects After Angiotensin Converting Enzyme Inhibition
Brief Title: Increased Renal Oxygenation and Angiotensin Converting Enzyme Inhibition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Maria Antonieta Moraes, Doctorate, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4111/08
Record Dates: First submitted 2012-01-16; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Renal Disease
Keywords: ECA; BOLD-MRI; kidney
MeSH Terms: conditions — Kidney Diseases | interventions — Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Captopril 25mg (Other): To study the renal blood oxygenation, the subjects took captopril (25mg).
  Interventions: Drug: captopril 25mg

INTERVENTIONS:
Drug: captopril 25mg — renal blood oxygenation after captopril
  Other Names: BOLD-MRI

SUMMARY:
It is well established that renal hypoxia is associated with the development of renal injury. The purpose of this study is measure the alterations in renal blood oxygenation after angiotensin II converting enzyme inhibition. The understanding of kidney adaptive mechanisms to renin angiotensin system effects in healthy subjects will be useful for the early detection of renal disease and for the development of new therapies to decrease the progression of the disease and its consequences.

DETAILED DESCRIPTION:
Subjects The study will be conducted under a protocol (number 4111/08) approved by the Ethics Committee of the Instituto de Cardiologia do Rio Grande do Sul-Fundação Universitária de Cardiologia/Brazil. After giving their informed consent,the patients will participate in the study. None of the subjects will take medication,food and water overnight. All measurements will be performed at the end of the morning.

After control BOLD-MRI measurements acquisition, subjects will take an oral ACE inhibitor (captopril 25 mg). Thirty minutes after captopril administration, without moving from the scanner, blood pressure will be measured and a second BOLD acquisition will be performed to detect a possible alteration in the renal oxygenation. Data will be collected by two radiologists and interpreted by a physician and a physiologist.

MR Imaging Technique Images were acquired using 1.5T HDx (Sigma, GE Healthcare, Waukesha, Win) and an 8 channels body coil.

Localizer images will be performed with axial and sagittal planes following the long axis of both kidneys, using breath hold and fast spoiled gradient echo (FSPGR) technique.

Oblique axial and coronal reference images will be acquired for color maps following approximately the short and long axis of both kidneys using FSPGR with the following parameters: FOV=40cm, matrix 256x128, slice thickness=5cm, slice gap 6cm, 3 slices per plane in one breath hold. TR=150ms, TE=min full, FLIP=90, rBW=62KHz, 1NEX. This sequence provides an excellent contrast between cortex and medulla and avoid the unnecessary use of a contrast agents.

BOLD sensitive images will be acquired using the multiple echo FGRE sequence with the same geometrical parameters. The reference images considered will have the following parameters: TR = 60ms, FLIP=30, rBW=60KHz, 16 echoes from TE=2.1ms until 49.6ms, echo interval of 3.2ms, 1 NEX.

BOLD imaging Data Processing Bold image processing will be performed using the Function R2* module for R2*/T2* fitting, assuming single exponential decay without constant offset at AW4.3 (GE Healthcare).

For visualization and quantification, R2* parametric maps will be generated for each slice.(11, 18-19) A Puh Talium color table will be used, since it was a dynamic range with minimum value set at 7.0/sec and maximum value at 23/sec. Color will be ranged from blue to red, close to minimum R2* and below and close to maximum R2* and above, respectively. The green/yellow will be assumed as intermediate. When a position mismatch due to a different breath hold state, anatomical fat suppressed FSPGR images were used as transparent references over a parametric map or original BOLD images.

One slice out of three, which provided the best differentiation between cortex and medulla and minimum partial volume, will be selected for quantification. A total of 6 regions of interest (ROI) with a 9 pixel size were used, 3 positioned at the cortex and 3 at the medulla for each plane.

The ROIs will be positioned at the cortex according to the anatomical reference image (light gray) and blue on the parametric map. The ROIs will be positioned at the medulla using either the anatomical reference image (dark gray) or the parametric map that showed a green, yellow and red gradient (figure 1). Areas with susceptibility artifacts, such as bowel gas or areas with renal hilum vessels, will be avoided.

Data analysis The statistical analysis will be determined by variance test for three repeated measures (ANOVA). Data are presented as the mean ± SD. P<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* healthy female between 45 and 55 years

Exclusion Criteria

* man and
* health female below 45 and above 55 years

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Measure the renal blood oxigenation after angiotensin converting enzyme inhibition | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MAntonieta Moraes, Dr, Study Chair — Instituto de Cardiologia do Rio Grande do Sul

REFERENCES:
- [Derived] Stein A, Goldmeier S, Voltolini S, Setogutti E, Feldman C, Figueiredo E, Eick R, Irigoyen M, Rigatto K. Renal oxygen content is increased in healthy subjects after angiotensin-converting enzyme inhibition. Clinics (Sao Paulo). 2012 Jul;67(7):761-5. doi: 10.6061/clinics/2012(07)10. PMID 22892920